CLINICAL TRIAL: NCT00100399
Title: A Randomized, Double-blinded, Placebo Controlled Phase III Study to Evaluate the Immunogenicity and Safety of GSK Bio Influenza Vaccine (Fluarix) Administered Intramuscularly in Healthy Adults
Brief Title: Fluarix Immunogenicity and Safety Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 04-098; 104233
Record Dates: First submitted 2004-12-30; First posted 2004-12-31 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2007-03

CONDITIONS: Influenza
Keywords: influenza, flu, Fluarix, vaccine, GSK, immunogenicity
MeSH Terms: conditions — Influenza, Human | interventions — fluarix

INTERVENTIONS:
Biological: Fluarix

SUMMARY:
The purpose of this study is to test the immune response caused by investigational Fluarix vaccine in healthy people aged between 18-64 years in the U.S.A. Up to 1050 volunteers at 4 centers will receive Fluarix or Placebo (saline), and their responses will then be compared. Subjects will be placed by age into 2 groups (18 to 49 years old and 50 to 64 years old), then randomly assigned to receive a dose of Fluarix or Placebo by injection into a muscle. There will be 2 phases in this study: (1) the active study phase (2 visits) for all subjects; and (2) the cross-over phase, only for subjects enrolled in the placebo group who accept to receive Fluarix. Blood samples will be obtained in order to measure immune response to the vaccine. On the day of vaccination, volunteers will receive a diary card to record information on symptoms experienced during the next 3 days. Subject participation in either group will be up to 2 months.

DETAILED DESCRIPTION:
This study is a randomized, double-blinded, placebo controlled Phase III study to evaluate the immunogenicity and the safety of GSK Bio influenza vaccine (Fluarix) administered intramuscularly in healthy adults aged 18 to 64 years. Vaccination is currently the most effective means of controlling influenza and preventing its complications and mortality in persons at risk. Following vaccination, seroprotective antibody titers are achieved in a high proportion of vaccinated subjects. GlaxoSmithKline Biologicals (GSK Bio) has been marketing an inactivated influenza split vaccine (Fluarix®) since 1992. More than 126 million doses have been distributed and the vaccine is registered in 78 countries. It has been well tolerated and has proven to be highly immunogenic when injected by the intramuscular route.

ELIGIBILITY:
Inclusion Criteria:

1. A male or female age between18-64 years at the time of the vaccination.
2. Subjects who the investigator believes can and will comply with the requirements of the protocol (e.g., return for follow-up visit and completion of the diary cards) should be enrolled in the study.
3. Written informed consent obtained from the subject.
4. Free of obvious health problems as established by medical history and clinical examination before entering into the study.
5. Female subjects must be of non-childbearing potential, i.e. either surgically sterilized or one year post-menopausal. If subject is of childbearing potential, she must be abstinent or have used adequate contraceptive precautions (e.g. intrauterine contraceptive device; oral contraceptives or other equivalent hormonal contraception, e.g. progestogen-only implantable, cutaneous hormonal patch or injectable contraceptives, diaphragm or condom in combination with contraceptive jelly, cream or foam) for 30 days prior to vaccination. She must also have a negative pregnancy test at study entry and must agree to continue such precautions for two months after completion of vaccination.

Exclusion Criteria:

1. Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the administration of the study vaccine, or planned use during the study period.
2. Has received any other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrollment in this study.
3. Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the administration of the study vaccine. (For corticosteroids, this will mean prednisone, or equivalent, >= 0.5 mg/kg/day.)
4. Any medically diagnosed or suspected immunodeficient condition based on medical history and physical examination (no laboratory testing required).
5. Administration of immunoglobulins and/or any blood products within the three months preceding the administration of the study vaccine or during the study.
6. History of hypersensitivity to a previous dose of influenza vaccine.
7. History of allergy or reactions likely to be exacerbated by any component of the vaccine including egg, chicken protein, formaldehyde, gentamicin sulfate or sodium deoxycholate.
8. Previous vaccination against influenza (2004-2005 influenza vaccine) within the 9 months prior to enrollment.
9. Acute disease at the time of enrollment. (Acute disease is defined as the presence of a moderate or severe illness with or without fever. All vaccines can be administered to persons with a minor illness such as diarrhea, mild upper respiratory infection with or without low-grade febrile illness, i.e. Oral temperature <37.5°C (99.5°F) / Axillary temperature <37.5°C (99.5°F)).
10. Acute clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
11. Major congenital defects or serious chronic illness.
12. History of any neurologic disorders, including history of Guillain Barré syndrome
13. History of seizures, with the exception of a single febrile seizure during childhood.
14. Pregnant or lactating female.
15. Female planning to become pregnant or planning to discontinue contraceptive precautions within 2 months of enrollment in this study.
16. Has an underlying medical condition for which influenza vaccination is recommended: chronic heart or lung conditions, including asthma; metabolic diseases; kidney disease; blood disorder (such as sickle cell anemia); weakened immune systems, including HIV/AIDS.
17. 18 years of age and on chronic aspirin therapy
18. Residents of nursing homes and long term care facilities.
19. Health care workers involved in direct patient care.
20. Out-of-home caregivers and household contacts of children <6 months.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1050
Dates: Start 2004-12; Study Completion 2004-12

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Maryland Baltimore, Baltimore, Maryland
  - University of Rochester, Rochester, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Baylor College of Medicine, Houston, Texas